CLINICAL TRIAL: NCT04220879
Title: Study on Intraocular Structural Parameters and Surgical Effect Before and After the Onset of Malignant Glaucoma
Acronym: MG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019KYPJ148
Record Dates: First submitted 2020-01-05; First posted 2020-01-07 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Glaucoma; Malignant Glaucoma
Keywords: Malignant Glaucoma; Biometric Measurements
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Malignant Glaucoma: To determine the biometric measurements.
- Fellow Eyes: To determine the biometric measurements.
- Matched Eyes: To determine the biometric measurements.

SUMMARY:
In this retrospective observational study, we collected intraocular structure parameters of malignant glaucoma and primary angle closure glaucoma. Anterior chamber depth (ACD) and width (ACW), lens vault (LV), ciliary process-ciliary process distance(CCD), trabecular-ciliary processes distance (TCPD), ciliary body max thickness (CBMT), peripheral iris thickness (PIT), trabecular ciliary process angle (TCPA), and anterior vault (AV), were measured by ultrasound biomicroscopy. Other parameters measured by A-scan ultrasonography and optical coherence tomography. To analyze the high risk factors and the possible pathogenesis of the disease and discuss the long-term effect of different treatment methods.

DETAILED DESCRIPTION:
Outcome Measures:

Anterior chamber depth (ACD) and width (ACW), lens vault (LV), ciliary process-ciliary process distance(CCD), trabecular-ciliary processes distance (TCPD), ciliary body max thickness (CBMT), peripheral iris thickness (PIT), trabecular ciliary process angle (TCPA), and anterior vault (AV), were measured by ultrasound biomicroscopy. Other parameters measured by A-scan ultrasonography and optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria: (1) history of operation, (2) diagnosis of MG, and (3) eyes with clear optical media.

Exclusion Criteria:(1)hypertension or diabetes and (2) diagnosis of ocular fundus diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients >=18 years old with or without malignant glaucoma
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-08-24 (Estimated); Study Completion 2020-11-24 (Estimated)

PRIMARY OUTCOMES:
Trabecular ciliary process angle | baseline
  TCPA is measured with its apex at the scleral spur, one arm along the posterior corneal surface, and another arm along the most anterior surface of the ciliary body
Choroidal vascularity parameter | baseline
  Choroidal vascularity parameter is a vessel ratio measured by optical coherence tomographic images

CONTACTS AND LOCATIONS:
Overall Officials: Chengguo O Zuo, Study Director — Zhognshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) needed to be keep security.